CLINICAL TRIAL: NCT01396603
Title: Pilot Study to Evaluate Optical Frequency Domain Imaging for Diagnosis of Central Airway Disease
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Melissa J. Suter, Assistant Professor of Medicine, Massachusetts General Hospital
Other Study IDs: 2008P001254; R00CA134920 (NIH)
Record Dates: First submitted 2011-07-15; First posted 2011-07-19 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Squamous Cell Lung Cancer; Lung Cancer
Keywords: Optical Frequency Domain Imaging; Optical Coherence Tomography; Optical biopsy; Comprehensive Microscopy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will evaluate a new imaging technology, termed optical frequency domain imaging (OFDI) for detecting and diagnosing pulmonary malignancy in the central airways.

DETAILED DESCRIPTION:
The prevalence and high mortality rate associated with lung squamous cell carcinoma and the lack of any widely accepted screening and surveillance tools, highlights the need for new imaging paradigms that will ultimately lead to a reduction in patient mortality.

Bronchial carcinoma-in-situ will progress to invasive cancer in over 40% of individuals, and although the progression occurs over a long period of time, the majority of carcinomas are detected in the later stages of disease development, offering patients only a slim chance of cure. Although significant effort in the development of screening paradigms for the detection of lung cancer in the central airways have been made, to date there is still no widely accepted and validated approach. Optical frequency domain imaging (OFDI) is a recent derivative of optical coherence tomography (OCT). OFDI can be used to conduct volumetric microscopy of the airways at a resolution comparable with architectural histopathology. The long term goal of this study is to use OFDI to screen the airways with the hope of detecting squamous cell carcinoma at an early more curable stage.

Standard of care bronchoscopy preparation and procedures will be followed including moderate sedation, pulse oximetry and blood pressure monitoring as per department protocol. A combination of currently approved bronchoscopy techniques including standard white light bronchoscopy, autofluorescence bronchoscopy, and narrow band imaging will be used to assess the airways. Bronchial regions of interest (ROI) suspected to be premalignant or malignant, will be imaged using the OFDI system and catheter prior to biopsy acquisition. It is anticipated that a minimum of 3 OFDI-biopsy correlated pairs from each study participant will be obtained. An additional OFDI and biopsy will be obtained from a normal ROI. It is expected that the experimental procedure will add less than 10 minutes to the total length of the bronchoscopy procedure, but a stopping rule will be instituted to ensure that the experimental procedure does not exceed 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bronchoscopy for known or suspected pulmonary malignancy in the central airways
* Patients must be over the age of 18
* Patient must be able to give informed consent
* Women with child bearing potential must have a negative pregnancy test the day before or the day of the procedure.

Exclusion Criteria:

- Patient does not meet the requirements to undergo clinical bronchoscopy, as determined by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for bronchoscopy procedures in the Pulmonary and Critical Care Department at Massachusetts General Hospital for the evaluation of known or suspected pulmonary malignancy will be enrolled in this study. Study patients will receive standard of care for pulmonary disease consistent with national guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of imaging device | on going

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Suter, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States